CLINICAL TRIAL: NCT05259709
Title: A First-in-Human Study of 89Zr-DFO-REGN5054 (Anti-CD8) Positron Emission Tomography in Patients With Solid Malignancies Treated With Cemiplimab
Brief Title: A Study of ImmunoPet Imaging Using 89Zr-DFO-REGN5054 in Adult Participants With Solid Cancers Treated With Cemiplimab
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5054-ONC-1843; 2019-001604-38 (EudraCT Number); 2024-515351-37-00 (EU CTIS Number)
Record Dates: First submitted 2022-01-24; First posted 2022-02-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Positron Emission Tomography (PET) scan; Immuno-PET
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single ascending dose of 89Zr˗DFO˗REGN5054 followed by fixed dose of cemiplimab (Experimental): Part A:
  Doses of 89Zr˗DFO˗REGN5054 may be reduced based upon assessment.
  Interventions: Drug: 89Zr˗DFO˗REGN5054; Drug: cemiplimab
- Defined dose of 89Zr˗DFO˗REGN5054 followed by fixed dose of cemiplimab (Experimental): Part B:
  Defined dose of 89Zr˗DFO˗REGN5054 determined in Part A.
  Interventions: Drug: 89Zr˗DFO˗REGN5054; Drug: cemiplimab

INTERVENTIONS:
Drug: 89Zr˗DFO˗REGN5054 — Administered by intravenous (IV) infusion during Part A and B.
Drug: cemiplimab — Administered by IV infusion every 3 weeks (Q3W).
  Other Names: REGN2810; Libtayo

SUMMARY:
This study is researching an experimental drug called 89Zr-DFO-REGN5054 and cemiplimab. The study is focused on patients with a type of cancer that can be potentially imaged using 89Zr-DFO-REGN5054 and show special tumor features that may be important to the way the immune system fights cancer.

The aim of the study is to study the safety and tolerability (how the body reacts to the drug) of the imaging agent 89Zr-DFO REGN5054.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drugs (which could make the study drugs less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

* Advanced or metastatic solid tumors that may respond to anti-programmed cell death 1 (PD-1) immunotherapy
* Measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Adequate organ and bone marrow function as defined in the protocol
* Willing and able to comply with clinic visits and study-related procedures (including required tumor biopsy for Part B)

Key Exclusion Criteria:

* Currently receiving another cancer treatment or inadequate time since last therapy, as defined in the protocol
* Has not yet recovered from acute toxicities from prior therapy; exceptions defined in the protocol
* Prior treatment with a blocker of the PD-1/Programmed death ligand 1 (PD-L1) pathway
* Currently receiving or has received chimeric antigen receptor (CAR-T) cell therapy
* Symptomatic or untreated brain metastases, leptomeningeal disease, or spinal cord compression
* Known history of or any evidence of interstitial lung disease, active, noninfectious pneumonitis (past 5 years) or active tuberculosis

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Up to day 8, after the infusion of 89Zr˗DFO˗REGN5054
  Part A
Incidence and severity of TEAEs | Up to approximately week 115
  Part A and B

SECONDARY OUTCOMES:
Clinical dosimetry based on tissue radiation absorbed dose calculated from positron emission tomography (PET) image acquisition data | On days 1, 5 and 8
  After injection of 37 megabecquerel (MBq) of 89Zr-DFO-REGN5054, a series of whole-body positron emission tomography (PET) images will be obtained over a period of up to 8 days and corrected for attenuation by low-dose computed tomography (CT) scans using PET/CT. The radiation effective dose per organ/tissue will be calculated for each organ using Organ Level INternal Dose Assessment/EXponential Modeling (OLINDA/EXM). The unit of effective dose per organ/tissue will be millisievert per Minimum Base Quantity (MBq) for each participant's organ/tissue. The final values for each organ will be averaged across participants for each mass dose
Clinical dosimetry based on tissue radiation effective dose calculated from PET image acquisition data | On days 1, 5 and 8
  After injection of 37 MBq of 89Zr-DFO-REGN5054, a series of whole-body PET images will be obtained over a period of up to 8 days and corrected for attenuation by low-dose CT scans using PET/CT. The radiation effective dose for the whole body will be calculated using OLINDA/EXM software. The unit of effective dose will be millisievert per MBq for the whole body for each participant. The final values will be averaged across participants for each mass dose.
Concentration of 89Zr-DFO-REGN5054 in serum | On days 1, 5 and 8
  Part A
Serum imaging agent activity concentration of area under the curve (AUC0-7) | Up to day 8
  Part A
89Zr-DFO-REGN5054 uptake across cluster of differentiation 8 (CD8)-expressing normal tissues and tumors | At the time of imaging, up to day 8
  Part A and Part B
Blood pool uptake of 89Zr-DFO-REGN5054 with subsequent calculation of standardized uptake value (SUV) tumor-to-blood ratios | At the time of imaging, up to day 8
  Part A and Part B
Association of 89Zr˗DFO˗REGN5054 autoradiographic signal intensity distribution with CD8 expression in tumor tissues | At Baseline
  Part A and Part B
Association of 89Zr-DFO-REGN5054 uptake with CD8 expression in tumor tissues | At Baseline
  Part B
Association of tumor-to-blood ratio of 89Zr-DFO-REGN5054 with CD8 expression in tumor tissues | At Baseline
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/